CLINICAL TRIAL: NCT02365259
Title: Effect of UVB Phototherapy on Serum Vitamin D in Persons With Multiple Sclerosis; a Placebo Controlled Study
Brief Title: Phototherapy in Persons With Multiple Sclerosis
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Illinois at Urbana-Champaign (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 15178
Record Dates: First submitted 2015-02-02; First posted 2015-02-18 (Estimated); Last update posted 2015-02-18 (Estimated); Status verified 2015-02

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Phototherapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Phototherapy (Experimental): This arm involves exposure to a UVB phototherapy device 3 times per week over 8 weeks.
  Interventions: Device: Phototherapy
- Shame phototherapy (Placebo Comparator): This arm is identical with experimental arm, except that participants will be exposed to non-UVB florescent light.
  Interventions: Device: Phototherapy

INTERVENTIONS:
Device: Phototherapy — Participants will be exposed to phototherapy according to the 2014 Guidelines issued by the American Academy of Dermatology 3 days per week over an 8-week period.

SUMMARY:
The current study examines the effect of phototherapy equipped with Narrow Band UVB lamps on vitamin D production in persons with MS.

DETAILED DESCRIPTION:
Participants will be exposed to phototherapy according to the 2014 Guidelines issued by the American Academy of Dermatology 3 days per week over an 8-week period.

ELIGIBILITY:
Inclusion Criteria:

* Female with multiple sclerosis

Exclusion Criteria:

* Inability to stand still in a stabilized fashion without risk of falling for up to 6 minutes
* Known medical history of calcium disorder or knowledge of high calcium levels
* Known medical history of hyper-parathyroidism
* Current supplementation with oral vitamin D
* Known allergy to vitamin D
* History of cancer of any type including but not limited to skin cancer
* Obesity defined as BMI > 30
* Known history of fat malabsorption conditions (i.e., steatorrhea)
* Current use of anti-epileptic medication
* Current use of glucocorticoids
* Fitzpatrick skin types I and VI using the Fitzpatrick skin type analysis
* Recent use of tanning facilities

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2015-01; Primary Completion 2016-02 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Serum Vitamin D at 4 and 8 weeks | 0, 4, and 8 weeks
  Venous blood will be collected to quantify levels of circulating Vitamin D.

SECONDARY OUTCOMES:
Change from Baseline in Walking Speed at 4 and 8 weeks | 0, 4, and 8 weeks
  Participants will walking for 25-feet as fast, but safely, as possible on an instrumented gait mat for measuring gait speed.
Change from Baseline in Cognitive Function at 4 and 8 weeks | 0, 4, and 8 weeks
  Participants will complete neuropsychological assessments of processing speed and learning and memory.
Change from Baseline in Mood State at 4 and 8 weeks | 0, 4, and 8 weeks
  Participants will complete a 30-item self-report measure of overall mood.

CONTACTS AND LOCATIONS:
Overall Officials: Robert W Motl, PhD, Principal Investigator — University of Illinois at Urbana-Champaign
Locations (1):
- Exercise Neuroscience Research Laboratory, Urbana, Illinois, United States